CLINICAL TRIAL: NCT04934046
Title: Clinical Evaluation of a New Multipurpose Whole-body CZT Camera in DaTSCAN Brain Scintigraphy: a Head-to-head Comparison With a Conventional System.
Brief Title: Evaluation of Dopaminergic Denervation by DaTSCAN Brain Scintigraphy Using a New Multipurpose CZT System
Acronym: STARDAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As the team at Nancy University Hospital published the same study last year, on the competing CZT 3D system (Veriton), our study is no longer relevant.
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRO-2020-21
Record Dates: First submitted 2021-03-09; First posted 2021-06-22 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
Keywords: DaTSCAN; Multipurpose CZT camera
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: All patients will undergo SPECT acquisitions with both new multipurpose CZT camera and conventional SPECT camera.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaTSCAN brain scan images from the new CZT SPECT system (Experimental): All patients will undergo additional SPECT acquisition (30min added time approximately), with no added radiation, with both new multipurpose CZT camera (StarGuide system, GE Healthcare, Haïfa, Israel) and conventional SPECT camera (Discovery 670, GE Healthcare, Haïfa, Israel)
  Interventions: Other: Additional acquisition

INTERVENTIONS:
Other: Additional acquisition — Additional SPECT acquisition (30min added time approximately), with no added radiation

SUMMARY:
DaTSCAN is an important tool in the diagnosis and clinical management of Parkinson's syndromes.

New cadmium-zinc-telluride (CZT) systems allow time and/or dose reduction. This can be interesting in DaTSCAN acquisitions as those are long-lasting, often on difficult patients.

This study will evaluate the diagnostic performances of a new 3D-ring CZT camera in DaTSCAN SPECT.

DETAILED DESCRIPTION:
DaTSCAN is an important tool in the diagnosis and clinical management of Parkinson's syndromes, particularly for the diagnosis of Parkinson's disease or in the exploration of dementia-type neurodegenerative diseases.

The acquisition of tomoscintigraphic images is performed 3 hours after injection and lasts approximately 30 minutes on a conventional gamma camera.

Recently, the introduction of systems equipped with cadmium-zinc-telluride (CZT) technology has made it possible to reduce acquisition times and/or injected doses. Among these systems, some new 3D-ring CZT cameras allow tomoscintigraphic acquisitions to be carried out from the outset for the exploration of different organs.

Patients included in this study will be double scanned both on a conventional camera and on the new multipurpose CZT system, with CT.

The primary objective is to evaluate the diagnostic concordance between the DaTSCAN brain scintigraphy images from the new CZT SPECT/CT system and those from the conventional SPECT camera, when visually interpreted blindly by experienced observers (nuclear medicine physicians), according to a diagnostic scale.

Striatal binding ratios (SBR) will also be compared. Time reduction will also be evaluated on DaTSCAN SPECT data from the new multi-purpose CZT system.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to our Nuclear Medicine department for DaTSCAN scintigraphy.

Exclusion Criteria:

* Under 18 years-old patients.
* Pregnant women or at risk of pregnancy.
* Breast feeding.
* Painful patients.
* Patients under guardianship.
* Patients in whom a standard examination is not feasible (agitation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Change in the visual Benamer Scale between new and conventional SPECT systems | Day 0
  Evaluation will be made by an experienced observer (senior physician of the nuclear medicine department), for images obtained for each of the patients included, according to the Benamer's 5-category scale with 5 categories (normal, reduce type1, reduce type 2, reduce type 3, other reductions)

SECONDARY OUTCOMES:
Change in the Striatal Binding ratios (defined as ratio between striatal uptake and background uptake) between new and conventional SPECT systems | Day 0
  SBR obtained with each of the 2 methods, at the end of the optimal image acquisition time and at reduced time.
Evaluation of time reduction. | Day 0
  Visual diagnostic classification of scintigraphic images on the Benamer scale when reducing the acquisition time, for each of the 2 acquisition methods.
Evaluation of time reduction | Day 0
  visual diagnostic classification of scintigraphic images made by an experienced observer (senior physician of the nuclear medicine department), for the images obtained with each of the 2 scintigraphic methods used, for each of the patients included, on the simplified Benamer diagnostic scale with only 2 categories (category 1: normal images / other categories: abnormal images), at the end of the optimal time foreseen for the acquisition of the images as well as at reduced time.

CONTACTS AND LOCATIONS:
Overall Officials: Mattieu BAILLY, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR d'Orleans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benamer TS, Patterson J, Grosset DG, Booij J, de Bruin K, van Royen E, Speelman JD, Horstink MH, Sips HJ, Dierckx RA, Versijpt J, Decoo D, Van Der Linden C, Hadley DM, Doder M, Lees AJ, Costa DC, Gacinovic S, Oertel WH, Pogarell O, Hoeffken H, Joseph K, Tatsch K, Schwarz J, Ries V. Accurate differentiation of parkinsonism and essential tremor using visual assessment of [123I]-FP-CIT SPECT imaging: the [123I]-FP-CIT study group. Mov Disord. 2000 May;15(3):503-10. PMID 10830416
- [Background] Suwijn SR, van Boheemen CJ, de Haan RJ, Tissingh G, Booij J, de Bie RM. The diagnostic accuracy of dopamine transporter SPECT imaging to detect nigrostriatal cell loss in patients with Parkinson's disease or clinically uncertain parkinsonism: a systematic review. EJNMMI Res. 2015 Mar 17;5:12. doi: 10.1186/s13550-015-0087-1. eCollection 2015. PMID 25853018
- [Background] Kupsch AR, Bajaj N, Weiland F, Tartaglione A, Klutmann S, Buitendyk M, Sherwin P, Tate A, Grachev ID. Impact of DaTscan SPECT imaging on clinical management, diagnosis, confidence of diagnosis, quality of life, health resource use and safety in patients with clinically uncertain parkinsonian syndromes: a prospective 1-year follow-up of an open-label controlled study. J Neurol Neurosurg Psychiatry. 2012 Jun;83(6):620-8. doi: 10.1136/jnnp-2011-301695. Epub 2012 Apr 6. PMID 22492213
- [Background] Tolosa E, Borght TV, Moreno E; DaTSCAN Clinically Uncertain Parkinsonian Syndromes Study Group. Accuracy of DaTSCAN (123I-Ioflupane) SPECT in diagnosis of patients with clinically uncertain parkinsonism: 2-year follow-up of an open-label study. Mov Disord. 2007 Dec;22(16):2346-51. doi: 10.1002/mds.21710. PMID 17914722
- [Background] Djang DS, Janssen MJ, Bohnen N, Booij J, Henderson TA, Herholz K, Minoshima S, Rowe CC, Sabri O, Seibyl J, Van Berckel BN, Wanner M. SNM practice guideline for dopamine transporter imaging with 123I-ioflupane SPECT 1.0. J Nucl Med. 2012 Jan;53(1):154-63. doi: 10.2967/jnumed.111.100784. Epub 2011 Dec 8. No abstract available. PMID 22159160